CLINICAL TRIAL: NCT07275502
Title: Prospective Development and Validation of an Objective Classification for Difficult Facemask Ventilation: the MASCAN Score - Secondary Analysis of the Prospective Observational MASCAN Study
Brief Title: Prospective Development and Validation of an Objective Classification for Difficult Facemask Ventilation: the MASCAN Score
Status: Active, not recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-300636-WF
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Airway Management; Mask Ventilation; Noninvasive Ventilation
Keywords: Difficult facemask ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Difficult facemask ventilation remains poorly classified. Existing definitions rely on expert opinion and subjective rating of surrogates. This lack of standardization has led to highly variable reported incidences and inconsistencies in clinical practice and research.

This secondary analysis of the prospective observational MASCAN study aims to develop and validate a data-driven objective classification system for difficult facemask ventilation and to determine its diagnostic performance and calibration. Facemask ventilation was facilitated after anaesthesia induction in all patients. An independent observer systematically assessed potential indicators for difficult facemask ventilation that serve as candidate predictor variables for the fitting of a diagnostic multivariable logistic regression model and simplified score to classify difficult facemask ventilation. Cross-validated LASSO regression will be used for variable selection. The area under the receiver operating characteristic curve (AUROC) and calibration curves will be used to quantify the diagnostic performance and calibration, and optimal decision thresholds will be defined.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduling for ENT or OMS surgery in general anaesthesia, who require facemask ventilation and tracheal intubation after induction of anesthesia
* Patients aged at least 18 years
* Ability to understand the patient information and to personally sign and date the informed consent to participate in the study
* The patient is co-operative and available for the entire study
* Provided informed consent/patient representative

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Rapid sequence induction or other contraindications for facemask ventilation
* Planned awake tracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive sampling: Adult patients that undergo ENT or OMS surgery in a tertiary care hospital who require facemask ventilation and tracheal intubation after induction of anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Difficult facemask ventilation | 1 hour
  Alert documented in patients' health records by the airway operator following facemask ventilation (y/n)

SECONDARY OUTCOMES:
Impossible facemask ventilation | 1 hour
  Observed impossible facemask ventilation after induction of anaesthesia (y/n)
Airway-related adverse events | 1 hour
  Laryngospasm, bronchospasm, larynx trauma, airway trauma, soft tissue trauma, oral bleeding, edema, dental damage, corticosteroid application, accidental esophageal intubation, aspiration, hypotension or hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Principal Investigator — University Medical Centre Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology, Center for Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany